CLINICAL TRIAL: NCT02047149
Title: Phase I Study to Evaluate the Safety of Zileuton (Zyflo®) in Combination With Dasatinib (Sprycel®) in Patients With Chronic Myelogenous Leukemia
Brief Title: Evaluating the Safety of Zileuton (Zyflo®) in Combination With Dasatinib (Sprycel®) in Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jan Cerny, MD, PhD, Assistant Professor, Medicine, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA 180-338
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid | interventions — zileuton; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zileuton/Dasatinib (Experimental): zileuton/dasatinib: This is a traditional phase I design. Three dose levels of daily zileuton will be studied in conjunction with dasatinib to define the MTD
  Interventions: Drug: Zileuton (Zyflo®) Dasatinib (Sprycel®); Drug: Dosing with Zileuton/Dasatinib in CML; Drug: Daily dosing of Zileuton/Dasatinib; Drug: Daily dosing with Zileuton/Dasatinib for CML

INTERVENTIONS:
Drug: Zileuton (Zyflo®) Dasatinib (Sprycel®) — To determine the maximum dose of zileuton/dasatinib in subjects with CML
Drug: Dosing with Zileuton/Dasatinib in CML — Three dose levels of daily zileuton will be studied in conjunction with dasatinib to define the MTD
  Other Names: Zyflo® + Sprycel®
Drug: Daily dosing of Zileuton/Dasatinib — Three dose levels of daily zileuton will be studied in conjunction with dasatinib to define the MTD
  Other Names: Zyflo® + Sprycel®
Drug: Daily dosing with Zileuton/Dasatinib for CML — Three dose levels of daily zileuton will be studied in conjunction with dasatinib to define the MTD
  Other Names: Zyflo®; Sprycel®

SUMMARY:
Prospective nonrandomized phase I study

The purpose of this study is to determine safety and efficacy of zileuton when added to dasatinib in patients with chronic myelogenous leukemia (CML).

DETAILED DESCRIPTION:
The standard treatment for chronic myelogenous leukemia is therapy with tyrosine kinase inhibitors (TKIs). This treatment can diminish the amount of disease to very low levels that only very sensitive and specialized techniques can measure; it does not, however, provide a cure.

Dr. Shaoguang Li and colleagues at University of Massachusetts have published a unique discovery that the arachidonate 5-lipoxygenase (5-LO) gene (Alox5) is a critical regulator for LSCs in BCR-ABL-induced CML (Chen Y et al. Loss of the Alox5 gene impairs leukemia stem cells and prevents chronic myeloid leukemia. Nature Genetics 41:783-792, 2009). In the absence of Alox5, BCR-ABL failed to induce CML in preclinical studies. While deficiency in Alox5 had no effect on normal hematopoiesis, impairment of the LSCs function through differentiation and cell division of CML LSCs was observed. This defect led to a depletion of LSCs and a failure of CML development. Treatment with a 5-LO inhibitor (zileuton) also impaired the function of LSCs and prolonged survival. These results demonstrate that a specific target gene can be found in cancer stem cells and its inhibition can completely inhibit the function of these stem cells. These findings provide an exciting opportunity to develop the first anti-cancer stem cell therapy for treating CML.

Patients who did not respond or did not tolerate two TKIs will be considered for this study.

ELIGIBILITY:
Inclusion Criteria:

Target Population:

1. Patients with CML with known inadequate response (as appropriate for their CML status) to TKIs or known resistance will be considered for this study

* Patients who are resistant or not responding adequately to dasatinib as a first line therapy, but are not able or eligible to receive other effective second line treatment can be considered for participation in the study.
* Age > 18 years
* ECOG performance status ≤ 2
* Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN)
* Hepatic enzymes (AST, ALT ) ≤ 1.5 times the institutional ULN
* Serum Na, K+, Mg2+, Phosphate and Ca2+>= Lower Limit of Normal (LLN)
* Serum Creatinine < 2.3 mg/dL
* PT, PTT all Grade 0-1 3) Ability to take oral medication 4) Concomitant Medications
* Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy 5) Age and Sex
* Women of childbearing potential and men of fathering potential must use an adequate method of contraception to avoid pregnancy throughout the study to minimize the risk of pregnancy

Exclusion Criteria:

1. Sex and Reproductive Status

   * Women of childbearing potential and men of fathering potential unable or unwilling to use an adequate method of contraception to avoid pregnancy throughout the study to minimize the risk of pregnancy
2. Target Population

   * Patients intolerant of dasatinib.
3. Medical History and Concurrent Diseases

   * History of active malignancy during the past 5 years with the exception of nonmetastatic treated skin cancer (e.g. basal or squamous cell carcinoma ) or stage 0 cervical carcinoma
   * Patients known to be HIV-positive
   * Patients with active, uncontrolled infections
   * Concurrent medical condition which may increase the risk of toxicity, including:
   * Pleural or pericardial effusion of any grade
   * Cardiac Conditions:
   * Uncontrolled angina, congestive heart failure or MI within (6 months)
   * Diagnosed congenital long QT syndrome
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
   * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
   * Severe cardiac dysfunction (NYHA classification III-IV)
   * Severe pulmonary disease
   * History of significant bleeding disorder unrelated to cancer
4. Physical and Laboratory Test Findings

   * Hepatic dysfunction (serum bilirubin ≥ 2 x ULN, and/or ALT ≥ 3 x ULN, and/or AST ≥ 3 x ULN)
   * Renal dysfunction (creatinine ≥ 200 μmol/l or 2.3 mg/dl)
   * Subjects with hypokalemia or hypomagnesemia that cannot be corrected prior to dasatinib administration
5. Allergies and Adverse Drug Reactions

   * Patients with known allergic reaction or intolerance to either dasatinib or zileuton
6. Prohibited Treatments and/or Therapies

   * Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including:
   * quinidine, procainamide, disopyramide
   * amiodarone, sotalol, ibutilide, dofetilide
   * erythromycin, clarithromycin
   * chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
   * cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
   * Patients requiring anticoagulation with Coumadin
7. Other Exclusion Criteria

   * Prisoners or subjects who are involuntarily incarcerated.
   * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose (MTD) of zileuton when added to dasatinib in patients with CML | 36 mos

SECONDARY OUTCOMES:
To assess the efficacy of zileuton combined with dasatinib in terms of: | 36 mos
  * 5-lipoxygenase (5-LO) blockade in patients
  * The rate of hematological response (where applicable)
  * The rate of complete cytogenetic response (where applicable)
  * The rate of major molecular response (where applicable)
  * Assessment of residual CML stem cells

CONTACTS AND LOCATIONS:
Overall Officials: Jan Cerny, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Chen Y, Hu Y, Zhang H, Peng C, Li S. Loss of the Alox5 gene impairs leukemia stem cells and prevents chronic myeloid leukemia. Nat Genet. 2009 Jul;41(7):783-92. doi: 10.1038/ng.389. Epub 2009 Jun 7. PMID 19503090
- [Background] Shah NP, Kantarjian HM, Kim DW, Rea D, Dorlhiac-Llacer PE, Milone JH, Vela-Ojeda J, Silver RT, Khoury HJ, Charbonnier A, Khoroshko N, Paquette RL, Deininger M, Collins RH, Otero I, Hughes T, Bleickardt E, Strauss L, Francis S, Hochhaus A. Intermittent target inhibition with dasatinib 100 mg once daily preserves efficacy and improves tolerability in imatinib-resistant and -intolerant chronic-phase chronic myeloid leukemia. J Clin Oncol. 2008 Jul 1;26(19):3204-12. doi: 10.1200/JCO.2007.14.9260. Epub 2008 Jun 9. PMID 18541900
- [Background] Daley GQ, Van Etten RA, Baltimore D. Induction of chronic myelogenous leukemia in mice by the P210bcr/abl gene of the Philadelphia chromosome. Science. 1990 Feb 16;247(4944):824-30. doi: 10.1126/science.2406902.
- See also: The Alox5 gene is a novel therapeutic target in cancer stem cells of chronic myeloid leukemia — http://www.ncbi.nlm.nih.gov/pubmed/19823023
- See also: Novel Therapeutic Agents Against Cancer Stem Cells of Chronic Myeloid Leukemia — http://www.eurekaselect.com/71277/article